CLINICAL TRIAL: NCT03182686
Title: A Phase 3 Randomized Study to Confirm the Efficacy of an Intra-Articular Injection of Ampion™ in Adults With Pain Due to Severe Osteoarthritis of the Knee
Brief Title: AP-003-C Study to Confirm the Efficacy of Ampion™ in Adults With Pain Due to Severe Osteoarthritis of the Knee
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ampio Pharmaceuticals. Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AP-003-C
Record Dates: First submitted 2017-06-06; First posted 2017-06-09 (Actual); Results first posted 2022-08-08 (Actual); Last update posted 2022-08-09 (Actual); Status verified 2022-08

CONDITIONS: Osteoarthritis, Knee; Knee Osteoarthritis; Knee Arthritis; Knee Pain Chronic
Keywords: osteoarthritis; osteoarthritis of the knee; OA; OAK; Kellgren Lawrence (KL)
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- AMPION™ 4 mL dose (Experimental): 4 mL injection of Ampion
  Interventions: Biological: 4 mL injection of Ampion
- Placebo 4 mL dose (Placebo Comparator): 4 mL injection of Placebo
  Interventions: Drug: 4 mL Injection of Placebo

INTERVENTIONS:
Biological: 4 mL injection of Ampion — 4 mL injection of Ampion
  Arms: AMPION™ 4 mL dose
Drug: 4 mL Injection of Placebo — 4 mL Injection of Placebo
  Other Names: 0.9% Saline
  Arms: Placebo 4 mL dose

SUMMARY:
This is a phase 3 randomized study to confirm the efficacy of an intra-articular injection of Ampion™ in adults with pain due to severe osteoarthritis of the knee.

DETAILED DESCRIPTION:
A Randomized Study to Confirm the Efficacy of an Intra-Articular Injection of Ampion™ in Adults With Pain Due to Severe Osteoarthritis of the Knee

There will be a 7-day screening period for each subject followed by a 12-week participation period.

The primary trial objective is to evaluate the clinical efficacy of Ampion using the Outcome Measures in Rheumatology Clinical Trials and Osteoarthritis Research Society International (OMERACT-OARSI) (using the Western Ontario and McMaster Universities Arthritis Index (WOMAC) 3.1 Index and Patient's Global Assessment as assessments).

The secondary trial objectives are to evaluate the safety of a single intra-articular injection (4 mL) of Ampion.

ELIGIBILITY:
Inclusion Criteria:

* Able to provide written informed consent to participate in the study;
* Willing and able to comply with all study requirements and instructions of the site study staff;
* Must be ambulatory;
* Study knee must have a clinical diagnosis of osteoarthritis (OA) supported by radiological evidence (Kellgren Lawrence Grade IV) which is assessed locally (x-rays within the past 6 months of screening are acceptable);
* Moderate to moderately-severe OA pain in the study knee (rating of at least 1.5 on the WOMAC A, 5-point Likert Pain Subscale);
* Moderate to moderately-severe OA function in the study knee (rating of at least 1.5 on the WOMAC C, 5-point Likert Function Subscale);
* WOMAC A, 5-point Likert pain subscale <1.5 in the contralateral knee;
* Ability to discontinue non-steroidal anti-inflammatory drug (NSAID) use at Screening visit and/or 72 hours prior to the Baseline visit and for the duration of the clinical study (low-dose aspirin (81 mg) is allowed during the study);
* No analgesia (including acetaminophen) taken 24 hours prior to an efficacy measure;
* No known clinically significant liver abnormality (e.g. cirrhosis, transplant, etc.).

Exclusion Criteria:

* As a result of medical review and screening investigation, the Principal Investigator considers the subject unfit for the study
* A history of allergic reactions to human albumin (reaction to non-human albumin such as egg albumin is not an exclusion criterion)
* A history of allergic reactions to excipients in 5% human albumin (N-acetyltryptophan, sodium caprylate)
* Presence of tense effusions
* Inflammatory or crystal arthropathies, acute fractures, history of aseptic necrosis or joint replacement in the affected knee, as assessed locally by the Principal Investigator
* Isolated patella femoral syndrome, also known as chondromalacia
* Any other disease or condition interfering with the free use and evaluation of the study knee for the duration of the trial (e.g. cancer, congenital defects, spine osteoarthritis)
* Major injury to the study knee within the 12 months prior to screening
* Severe hip osteoarthritis ipsilateral to the study knee
* Any pain that could interfere with the assessment of study knee pain (e.g. pain in any other part of the lower extremities, pain radiating to the knee)
* Any pharmacological or non-pharmacological treatment targeting OA started or changed during the 4 weeks prior to randomization or likely to be changed during the duration of the study
* Pregnancy or planning to become pregnant during the study
* Use of the following medications:

  1. No intra-articular (IA) injected medications in the study knee during the study (or 12 weeks prior to Baseline).
  2. No analgesics containing opioids.
  3. NSAIDs are not permitted during the study; acetaminophen is available as a rescue medication during the study from the provided supply.
  4. No topical treatment on the study knee during the study
  5. No significant anticoagulant therapy (e.g. Heparin or Lovenox) during the study (treatment such as low-dose Aspirin (81 mg) and Plavix are allowed)
  6. No systemic treatments that may interfere with safety or efficacy assessments during the study
  7. No immunosuppressants
  8. No use of systemic or intra-articular corticosteroids
* No human albumin treatment in the 3 months before randomization or throughout the duration of the study

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Actual)
Dates: Start 2017-06-19 (Actual); Primary Completion 2017-12-07 (Actual); Study Completion 2017-12-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Howard Levy, MD, Study Director — Ampio Pharmaceuticals. Inc.
Locations (13):
- United States (13):
  - Central Research Associates, Inc., Birmingham, Alabama
  - CORE Orthopaedic Medical Center, Encinitas, California
  - St. Joseph Heritage, Fullerton, California
  - Artemis Institute for Clinical Research, San Diego, California
  - Westlake Medical Research, Thousand Oaks, California
  - Drug Studies America, Marietta, Georgia
  - Healthcare Research Netword, Blue Island, Illinois
  - Heartland Research Associates, Wichita, Kansas
  - Arthritis Treatment Center, Frederick, Maryland
  - Healthcare Network Research, Hazelwood, Missouri
  - Coastal Carolina Center at Lowcountry Orthopaedics, North Charleston, South Carolina
  - Tekton Research, Austin, Texas
  - Northwest Clinical Research Center, Bellevue, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Salottolo K, Cole B, Bar-Or D. Intra-articular injection of the anti-inflammatory compound LMWF-5A in adults with severe osteoarthritis: a double-blind prospective randomized controlled multi-center safety and efficacy trial. Patient Saf Surg. 2018 Jun 18;12:11. doi: 10.1186/s13037-018-0158-0. eCollection 2018. PMID 29910837

RESULTS

PARTICIPANT FLOW:
Groups:
- Ampion 4 mL Dose: Ampion (<5 kilodalton (kDa) ultrafiltrate of 5% Human Serum Albumin (HSA)), solution, 4 mL, single intra-articular injection
  Ampion: Ampion (<5 kilodalton (kDa) ultrafiltrate of 5% HSA)
- Saline 4 mL Dose: Saline, solution, 4 mL, single intra-articular injection
  Saline: 0.9% sodium chloride
Period: Overall Study
Arm/Group | Ampion 4 mL Dose | Saline 4 mL Dose
Started | 144 | 24
Completed | 137 | 24
Not Completed | 7 | 0
Not completed — Lost to Follow-up | 2 | 0
Not completed — Adverse Event | 2 | 0
Not completed — Withdrawal by Subject | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ampion 4 mL Dose | Saline 4 mL Dose | Total
Number analyzed (Participants) | 144 | 24 | 168
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.74 (9.63) | 64.04 (6.25) | 62.92 (9.22)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 76 | 12 | 88
  Male | 68 | 12 | 80
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 1 | 6
  Not Hispanic or Latino | 139 | 23 | 162
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 3 | 1 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 27 | 6 | 33
  White | 111 | 16 | 127
  More than one race | 2 | 1 | 3
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 144 | 24 | 168
WOMAC Pain [Mean (Standard Deviation); unit: score on a scale] — The Western Ontario and McMaster Universities Arthritis Index (WOMAC) 3.1 evaluates Pain (5 items): during walking, using stairs, in bed, sitting or lying, and standing upright.
  Subjects respond to each subscale by using a 5-point Likert score. (0=none; 1=mild; 2=moderate; 3=severe; 4=extreme). Mean of the 5 scores constitutes the Baseline Pain Score.
  The minimum score on this scale is 0, and the maximum score is 4. Higher scores are indicative of higher levels of self-reported pain.
  score on a scale | 2.5 (0.56) | 2.4 (0.45) | 2.5 (0.55)
WOMAC Function [Mean (Standard Deviation); unit: score on a scale] — WOMAC 3.1 evaluates Physical Function (17 items): using stairs, rising from sitting, standing, bending, walking, getting in/out of a car, shopping, putting on/taking off socks, rising from bed, lying in bed, getting in/out of bath, sitting, getting on/off toilet, heavy/light domestic duties.
  Subjects respond to each by using a 5-point Likert score. (0=none; 1=mild; 2=moderate; 3=severe; 4=extreme). Mean of the 17 scores constitutes the Baseline Function Score. Minimum score is 0; maximum is 4.
  Higher scores indicate higher levels of limitations of self-reported physical function.
  score on a scale | 2.6 (0.53) | 2.5 (0.53) | 2.6 (0.53)
Patient's Global Assessment (PGA) [Mean (Standard Deviation); unit: score on a scale] — The Patient's Global Assessment of disease severity has subjects answer the following question: "Considering all the ways in which your arthritis affects you, please indicate how you are doing." Patients respond by using a 5-point Likert score (0=very well; 1=well; 2=fair; 3=poor; 4=very poor).
  Minimum score is 0; maximum is 4. Higher scores indicate greater patient's assessment of disease severity due to arthritis.
  score on a scale | 2.8 (0.80) | 2.7 (0.75) | 2.8 (0.79)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Classified as Responders
Description: Using the Outcome Measures in Rheumatology Clinical Trials and Osteoarthritis Research Society International (OMERACT-OARSI) criteria of WOMAC A Pain subscore, WOMAC C Function subscore, and PGA as composite endpoints. A patient in this study will be considered a responder for the purpose of efficacy analysis if the following criteria are met:
  (1) demonstration of ≥ 50% improvement AND a 1.0-unit change in pain OR 1.0-unit change in function OR
  If the patient does not meet this criterion, then the patient must demonstrate at least 2 of the following:
  * Improvement in pain (WOMAC A) ≥20% and a 0.5 point absolute change in pain from Baseline on the 5-point Likert scale
  * Improvement in function (WOMAC C) ≥20% and a 0.5 point absolute change in function from Baseline on the 5-point Likert scale
  * Improvement in patient global assessment (PGA) ≥20% and a 0.5 point absolute change in function from Baseline on the 5-point Likert scale
Time Frame: Determined from Baseline to 12 Weeks
Population: Intent to Treat (ITT)
Measure: Count of Participants; unit: Participants
Arm/Group | Ampion 4 mL Dose | Saline 4 mL Dose
Number analyzed (Participants) | 144 | 24
Participants | 102 | 15
Statistical Analysis 1: Comparison: Ampion 4 mL Dose vs Saline 4 mL Dose; H0:π ≤ π0 versus HA:π > π0 Where π0 is the hypothesized clinically significant value for the proportion of responders. The value will be 30% in this study. This test will be tested using an exact binomial test. That is, given the sample size of n, the number of responders X, and the value of π0 =0.30, then probability that X or more events would be observed will be calculated as the p-value. Since this is a one-sided test, the alpha level will be 0.025; Test type: Superiority; p < 0.0001, Fisher Exact

ADVERSE EVENTS:
Time Frame: 12 Weeks
Description: Patients will be followed for the occurrence of Adverse Events until 12 weeks after the first dose of study medication
Arm/Group | Ampion 4 mL Dose | Saline 4 mL Dose
All-Cause Mortality (participants affected / at risk) | 0/144 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/144 | 0/24
Other Adverse Events (participants affected / at risk) | 52/144 | 8/24
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ampion 4 mL Dose (N=144) | Saline 4 mL Dose (N=24)
Influenza-like illness (General disorders) | 0 | 1
Injection site joint pain (General disorders) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 1
Viral upper respiratory tract infection (Infections and infestations) | 4 | 0
Fall (Injury, poisoning and procedural complications) | 2 | 0
Procedural pain (Injury, poisoning and procedural complications) | 2 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 19 | 2
Arthropathy (Musculoskeletal and connective tissue disorders) | 2 | 0
Joint stiffness (Musculoskeletal and connective tissue disorders) | 3 | 2
Joint swelling (Musculoskeletal and connective tissue disorders) | 4 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 0
Synovial cyst (Musculoskeletal and connective tissue disorders) | 2 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 1
Headache (Nervous system disorders) | 4 | 0
Nausea (Gastrointestinal disorders) | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2017-11-09): https://cdn.clinicaltrials.gov/large-docs/86/NCT03182686/Prot_000.pdf
  • Statistical Analysis Plan (2017-11-14): https://cdn.clinicaltrials.gov/large-docs/86/NCT03182686/SAP_001.pdf